CLINICAL TRIAL: NCT03808792
Title: A Comparison Between Ultrasound, CT (CT) and Whole-body Diffusion-weighted MRI (WB-DWI/MRI) in the Assessment of Operability in Patients With Ovarian Cancer
Brief Title: Imaging Study in Advanced Ovarian Cancer
Acronym: ISAAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Ana Patrícia Pinto, Principal Investigator, Charles University, Czech Republic
Other Study IDs: č.j. 29/18
Record Dates: First submitted 2018-10-28; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Ultrasound; CT; WB-DW/MRI; Imaging
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer patients: Patients with abdominal or pelvic mass suspicious of primary ovarian, tubal or peritoneal cancer submitted to the index test (Ultrasound, CT and WB/DWI-MRI) with perspective of primary surgery
  Interventions: Diagnostic Test: Ultrasound, CT and WB-DWI/MRI

INTERVENTIONS:
Diagnostic Test: Ultrasound, CT and WB-DWI/MRI — Preoperative assessment with Ultrasound, CT and WB-DWI/MRI

SUMMARY:
The aim of the study is the assessment of tumour sites critical for the achievement of optimal cytoreduction in patients with advanced ovarian cancer using Ultrasound, CT and WB-DWI/MRI. The study uses an equivalence design with a hypothesis that cases with non-resectable disease identified by Index test (Ultrasound, CT and WB-DWI MRI) are equivalent to a portion of cases identified during surgery.

DETAILED DESCRIPTION:
Patients with abdominal or pelvic mass suspicious of primary ovarian, tubal or peritoneal cancer using subjective assessment by experienced sonographer (principal investigator) will be enrolled in the study and send to surgical planning. During surgical planning, the CT and MRI will be scheduled and the patient ́s consent will be requested if inclusion criteria are fulfilled. Please note, tumors with atypical morphology and/or tumor spread suspicious for secondary ovarian cancer will be first subjected to a tru-cut biopsy and will be included if histopathology confirms adnexal or peritoneal cancer.

Ultrasound will be always performed by the principal investigator in each center. Principal investigator is an ultrasound expert with level II or III EFSUMB accreditation (http://www.efsumb.org/). Operators performing ultrasound scan and radiologists performing CT or MRI will be well instructed and educated about standardized approach and criteria of inoperability. Sonographers and radiologists will be blinded to the results of other imaging modalities. If a patient already had CT or WB-DWI/MRI done by the referring hospital, the study radiologists will decide about the quality of imaging and necessity to repeat CT or WB-DWI/MRI.

The decision to treat by PDS (primary debulking surgery), or by NACT (neoadjuvant chemotherapy) with IDS (interval debulking surgery) will be based on departmental guidelines taking into account medical comorbidities and disease-related factors. If a patient is indicated for NACT a tru-cut biopsy or/and a diagnostic laparoscopy are performed. The clinicians will document why the primary debulking surgery was not considered. The surgery (laparoscopy, primary or interval debulking surgery) should always be performed within four weeks after the index test. Patients without surgical exploration will be excluded.

Surgeons performing laparoscopy will describe site to site involvement and in case of inoperability will take a biopsy and document reasons for abandoning laparotomy. In operable cases surgeons performing laparotomy will describe site to site involvement and where applicable reasons for not achieving optimal cytoreduction defined as no residual tumor left in situ at the end of surgery (R0).

If the patient has only ultrasound and CT (and not WB-DWI/MRI) she can still be included in the study. Similarly if the patient undergoes interval debulking surgery she can be included in the study if the index tests will be performed less than 4 week before IDS.

Clinical data and four evaluation forms will be filled in (Ultrasound, CT, MRI, Surgery) immediately after the procedure using electronic database. The evaluation form from histopathology will be filled when available by principal investigator. The database cannot be saved unless all the information required are filled in and it will not be available to any other investigator. Data will be submitted for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal or pelvic mass suspicious of primary ovarian, tubal or peritoneal cancer using subjective assessment by experienced sonographer.
2. Surgery (PDS or IDS) within 4 weeks from the index test.
3. 18 > Age < 80.
4. ECOG (Eastern Cooperative Oncology Group) grade < 3.
5. Patients after NACT can be included.

Exclusion Criteria:

1. Lesions suspected as being borderline ovarian tumors (BOT) on ultrasound.
2. Patients with supradiaphragmatic metastases
3. Contraindications to CT
4. Medical contraindications to surgery
5. Refusal or withdrawal of written informed consent
6. Time lapse between ultrasound and surgery more than 4 weeks
7. Current pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Study Population: Patients with an abdominal or pelvic mass suspicious of primary ovarian, tubal or peritoneal cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative identification of patients with ovarian/tubal cancer in whom optimal debulking (R0/R1) can not be achieved by US and CT scan. | 24 months
  Optimal debulking is defined as residual disease <1cm

SECONDARY OUTCOMES:
Assessment of the diagnostic performance in the detection of involvement of individual sites relevant for clinical management and in the detection of 24 individual sites described in the evaluation form. | 24 months
  1. Detection of involvement of individual sites relevant for clinical management:
     * Rectosigmoid
     * Colon (except ileocecum)
     * Ileocaecum
     * Lesser omentum
     * Small intestine
     * Liver
     * Diaphragm
     * Pleura
  2. Detection of 24 individual sites described in the evaluation form (17 peritoneal sites and 7 lymph nodes sites).
  The aim is to clarify the diagnostic performance of the different imaging methods in the assessment of tumor extent in form of peritoneal carcinomatosis and metastatic lymph nodes. The investigators want to establish the overall accuracy of each imaging modality in all the metastatic sites. The major interest lies in the sites that determine the extent of surgery and optimal cytoreduction, in particular bowel resection, lesser omentum, superficial liver metastases, diaphragm or pleura.
Prediction model of achievement of optimal cytoreduction. | 24 months
  Prediction of optimal cytoreduction based on preoperative imaging. Optimal cytoreduction is defined as no residual tumor left at the end of surgery (R0).
Markers influencing accuracy - FIGO stage | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods:
  FIGO stage - it will be analised if the accuracy of the imaging methods change between early stages (I-II) and late stages (III-IV) of the disease
Markers influencing accuracy - Histological type | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods:
  Histological type - it will be analised if the accuracy of the imaging methods change between serous type and other histological types
Markers influencing accuracy - Origin | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods: Origin - it will be analised if the accuracy of the imaging methods change between ovarian origin and tubal origin
Markers influencing accuracy - Intraperitoneal fluid | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods:
  Intraperitoenal fluid - it will be analised if the accuracy of the imaging methods change between < or = 400 mL and > 400 mL
Markers influencing accuracy - Age | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods:
  Age - it will be analised if the accuracy of the imaging methods change between women with < or = 65 and > 65 years old
Markers influencing accuracy - CA 125 | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods:
  CA 125 - it will be analised if the accuracy of the imaging methods change between < or = 300 U/mL and > 300 U/mL
Markers influencing accuracy - Postmenopausal status | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods:
  Postmenopausal status - it will be analised if the accuracy of the imaging methods change between premnopausal and postmenopausal status
Markers influencing accuracy - Body mass index | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods:
  Body mass índex - it will be analised if the accuracy of the imaging methods change between < or = 25 kg/m2 and > 25 kg/m2
Markers influencing accuracy - Image quality | 24 months
  Assessment of markers influencing diagnostic accuracy of individual methods:
  Image quality - it will be analised if the accuracy of the imaging methods change between good, moderate and poor image quality

OTHER OUTCOMES:
Patient Method Friendly Questionnaire | 24 months
  Evaluation of patients' experience of the imaging modalities using Patient Method Friendly Questionnaire.
  The aim of the questionnaire is to evaluate the overall experience through the different imaging methods and to evaluate relevant factors that may had a negative impact on the examination. The answers should be in a 4-point scale (1-very disappointing; 2-disappointing; 3- satisfied; 4-very satisfied) except the level of pain that should be in a 10-scale of pain (1 - no pain; 10 - maximum pain)
Excluded patients | 24 months
  Monitorization of excluded patients using an evaluation form filled by the principal investigator or study coordinator in each center. It has to be chosen one of the next options:
  1. Age <18 or > 80 years old
  2. Poor performance status ECOG >3
  3. Histologic report of biopsy of a non-gynecologic cancer
  4. Contraindications to upfront LPS or LPT (only tru-cut biopsy +/- NACT)
  5. Contraindications to CT
  6. Consent not given by the patient (denial or withdrawal of oral informed consent)
  7. Absence of insurance
  8. Time between ultrasound and surgery more than 4 weeks
  9. Current pregnancy
  10. Death
  11. Others, please specify:
Record of choice of treatment | 24 months
  Record of multidisciplinary team choice of primary surgery or neoadjuvant chemotherapy to clarify personal and external factors in decision making

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Fischerová, MD, PhD, Study Chair — Gynecologic Oncology Center, Department of Obstetrics and Gynecology, General University Hospital in Prague and 1st Medical Faculty of the Charles University, Prague, Czech Republic
Locations (1):
- Gynecologic Oncology Center in Prague, Prague, Czechia

REFERENCES:
- [Derived] Fischerova D, Pinto P, Pesta M, Blasko M, Moruzzi MC, Testa AC, Franchi D, Chiappa V, Alcazar JL, Wiesnerova M, Cibula D, Valentin L; collaborators. Ultrasound examiners' ability to describe ovarian cancer spread using preacquired ultrasound videoclips from a selected patient sample with high prevalence of cancer spread. Ultrasound Obstet Gynecol. 2025 May;65(5):641-652. doi: 10.1002/uog.29208. Epub 2025 Apr 18. PMID 40247746
- [Derived] Pinto P, Valentin L, Borcinova M, Wiesnerova M, Filip F, Burgetova A, Masek M, Lambert L, Chiappa V, Franchi D, Testa AC, Moro F, Avesani G, Panico C, Alessi S, Pricolo P, Vigorito R, Calareso G, Kocian R, Slama J, Fagotti A, Urbinati AMV, Signorelli M, Bertolina F, Cibula D, Fischerova D. Patient satisfaction with ultrasound, whole-body CT and whole-body diffusion-weighted MRI for pre-operative ovarian cancer staging: a multicenter prospective cross-sectional survey. Int J Gynecol Cancer. 2024 Jun 3;34(6):871-878. doi: 10.1136/ijgc-2023-005264. PMID 38531539